CLINICAL TRIAL: NCT04955184
Title: Comparing Cardiac Output Measurements Using a Wearable, Wireless, Non-invasive PPG-Based Device to a Swan Ganz Catheter During Ambulatory Assessment of CHF Patients
Brief Title: Comparing Cardiac Output Measurements Using a Wearable, Wireless, Non-invasive PPG-Based Device to a Swan Ganz Catheter
Status: Completed | Type: Observational
Sponsor: Biobeat Technologies Ltd. (Industry)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: CO-002-00
Record Dates: First submitted 2021-07-04; First posted 2021-07-08 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2021-12

CONDITIONS: Cardiac Output, Low; Cardiac Output, High; Congestive Heart Failure
Keywords: Non-Invasive Monitoring; Cardiac Output
MeSH Terms: conditions — Cardiac Output, Low; Cardiac Output, High; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: non-invasive monitoring — non-invasive measurements of cardiac output

SUMMARY:
Invasive pulmonary capillary wedge pressure measurements using a Swan-Ganz catheter (SGC) is considered the gold standard for cardiac output (CO) monitoring. In this prospective study, we will compare CO measurements between a PPG-based wearable monitor and a SGC in ambulatory CHF patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CHF

Exclusion Criteria:

* Pregnant women
* Pediatric patients
* Inability to sign an informed consent form

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients from both sexes with CHF arriving for an ambulatory assessment using a Swan-Ganz catheter in the Medical Center's Cath-lab.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-25 (Actual)

PRIMARY OUTCOMES:
Comparison of cardiac output obtained by a non-unvasive device to the invasive method | 2-4 hours per patient
  In each participant, a Swan-Ganz catheter will be inserted as part of their routine assessment, and cardiac output measurements will be compared with a non-invasive wearable and wireless PPG-based device.

CONTACTS AND LOCATIONS:
Overall Officials: Dean Nachman, MD, Principal Investigator — The Institute for Research in Military Medicine
Locations (1):
- The Hadassah Ein Kerem Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided
We aim to publish the results of this study in a peer-reviewed journal.

REFERENCES:
- [Derived] Nachman D, Eisenkraft A, Rahamim E, Ibrahimli M, Asenov A, Goldstein N, Kolben Y, Huly S, Ben Ishay A, Fons M, Tabi M, Merin R, Amir O, Asleh R. Assessing Cardiac Flow Measurements Using a Noninvasive Photoplethysmography-Based Device Compared to Invasive Pulmonary Artery Catheter. JACC Adv. 2025 Sep;4(9):102093. doi: 10.1016/j.jacadv.2025.102093. Epub 2025 Aug 22. PMID 40845743